CLINICAL TRIAL: NCT01652820
Title: Randomized Phase II Trial Using Concomitant Chemoradiation Plus Induction or Consolidation Chemotherapy for Unresectable Stage III Non-small Cell Lung Cancer Patients
Brief Title: Chemotherapy/Radiotherapy Versus Concomitant Chemotherapy Followed by Radiotherapy in Stage IIIB Non-small Cell Lung Cancer
Acronym: GECP0008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP 00-08 / TAX.ES1.209
Record Dates: First submitted 2012-07-17; First posted 2012-07-30 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non Small-cell Lung Cancer
Keywords: LUNG; DOCETAXEL; GEMCITABINE; CARBOPLATIN; RADIOTHERAPY
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel +Carboplatin +concomitant chemoradiation (Experimental): Docetaxel 20 mg/m2/weekly plus carboplatin AUC 2/weekly (first, docetaxel will be administered and after that, carboplatin will be administered) and concomitant chemoradiation (total dose of 60 Gy: 2 Gy/day, 5 days(week for 6 weeks)
  Interventions: Drug: Docetaxel 20mg/m2/week + carboplatin AUC 2/weekly - concomitant chemoradiation 2Gy/day; Drug: Docetaxel 40mg<7m2 d1,8, 21, 28+ gemcitabine 1200mg/m2 d1,8, 21, 28 + concomitant docetaxel 20mg/m2/w+carboplatin AUC 2/w+ concomitant RDT 2Gy/d
- C) Docetax+ gemcit +concom. docetax + carbopl. + RDT concom (Experimental): Docetaxel 40 mg/ m2 days 1, 8, 21 y 28 plus gemcitabine 1200 mg/ m2 days 1, 8, 21 y 28 followed by concomitant treatment Docetaxel 20 mg/m2/week plus carboplatin AUC 2/weekly and concomitant chemoradiation total dose of 60 Gy: 2 Gy/day, 5 days(week for 6 weeks)
  Interventions: Drug: Docetaxel 20mg/m2/week + carboplatin AUC 2/weekly - concomitant chemoradiation 2Gy/day; Drug: Docetaxel 40mg<7m2 d1,8, 21, 28+ gemcitabine 1200mg/m2 d1,8, 21, 28 + concomitant docetaxel 20mg/m2/w+carboplatin AUC 2/w+ concomitant RDT 2Gy/d

INTERVENTIONS:
Drug: Docetaxel 20mg/m2/week + carboplatin AUC 2/weekly - concomitant chemoradiation 2Gy/day
Drug: Docetaxel 40mg<7m2 d1,8, 21, 28+ gemcitabine 1200mg/m2 d1,8, 21, 28 + concomitant docetaxel 20mg/m2/w+carboplatin AUC 2/w+ concomitant RDT 2Gy/d

SUMMARY:
Randomized study in 2 arms, without any masking in patients with non small cell lung cancer, histologically or cytologically confirmed, not liable to surgery, stage IIIB or IIIA, according to the TNM classification of the American Joint Committee for cancer. In one arm will be administered concomitant radiotherapy and carboplatin-docetaxel-gemcitabine followed by docetaxel and, in the other arm will be administered docetaxel-gemcitabine followed by concurrent radiotherapy with carboplatin-docetaxel

ELIGIBILITY:
Inclusion Criteria:

* Unresectable stage IIIA or B NSCLC patients
* WHO PS 0 or 1
* Weight loss < 5 % within the last 3 months
* At least one measurable lesion
* Planning CT scan previous to randomization
* Written informed consent

Exclusion Criteria:

* Malignant effusion, supraclavicular node or SVCS
* PTV > 2000 cm3
* V20 > 35%
* FEV1 and DLCO both < 30% or 1 liter at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2001-10; Primary Completion 2006-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate | From enrollment to first response assesment
  The final response rates were 57% (arm B) and 56.9% (arm C). Arm A not available due to early closing

SECONDARY OUTCOMES:
Local control rate at 1 year | 1 year
Time to progression | From enrollment to first progression date
  Arm B: 7.6 months (m) and arm C: 9.2 m; p= 0.12)
Overall Survival | From enrollment to last follow up or death
  Arm B: 14.3 m and arm C: 14.7 m; p= 0.3

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Garrido, MD, Principal Investigator — Hospital Ramon y Cajal (Madrid); Rafael Rosell, MD, Principal Investigator — Germans Trias i Pujol Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrido P, Rosell R, Arellano A, Andreu F, Domine M, Perez-Casas A, Cardenal F, Arnaiz Mdel M, Moran T, Morera R, Isla D, Valencia J, Cobo M, Delgado R, Garcia-Gomez R, Calvo F, Zamora J, Ramos A, Massuti B. Randomized phase II trial of non-platinum induction or consolidation chemotherapy plus concomitant chemoradiation in stage III NSCLC patients: mature results of the Spanish Lung Cancer Group 0008 study. Lung Cancer. 2013 Jul;81(1):84-90. doi: 10.1016/j.lungcan.2013.03.009. Epub 2013 Apr 21. PMID 23611405